CLINICAL TRIAL: NCT00034892
Title: Efficacy and Tolerability of Olanzapine, Quetiapine and Risperidone in the Treatment of First Episode Psychosis: A Randomized Double Blind 52-Week Comparison
Brief Title: CAFE Comparison of Atypicals in First Episode of Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: University of North Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5077IL/0114
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Psychotic Disorders; Mental Health; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Psychological Well-Being; Mental Disorders | interventions — Olanzapine; Risperidone

INTERVENTIONS:
Drug: Olanzapine, risperidone

SUMMARY:
The purpose of this study is to compare the effectiveness, tolerability, and efficacy of the currently available atypical antipsychotic drugs olanzapine (2.5-20 mg/day), quetiapine (100-800 mg/day) and risperidone (0.5-4 mg/day) in patients with schizophrenia, schizophreniform disorder, or schizoaffective disorder who are experiencing their first psychotic episode.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet criteria for schizophreniform disorder, schizophrenia, or schizoaffective disorder with psychotic symptoms lasting 1-60 months
* Psychotic symptoms must have persisted at least one month, and not more thn 5 years (60 months)
* Patients must have no previous history of drug treatment (greater than a total of 16 weeks) with antipsychotics

Exclusion Criteria:

* Patients with history of psychotic disorder with recovery period of at least 3 months
* Female patients who are pregnant or nursing
* Patients with a known history of mental retardation

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (24):
  - Stanford, California
  - Miami, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Brooklyn, New York
  - New York, New York
  - Butner, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Kettering, Ohio
  - Philadelphia, Pennsylvania
  - Conroe, Texas
  - Research Site, Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Canada (2):
  - Calgary, Alberta
  - Halifax, Nova Scotia

REFERENCES:
- [Derived] Perkins DO, Gu H, Weiden PJ, McEvoy JP, Hamer RM, Lieberman JA; Comparison of Atypicals in First Episode study group. Predictors of treatment discontinuation and medication nonadherence in patients recovering from a first episode of schizophrenia, schizophreniform disorder, or schizoaffective disorder: a randomized, double-blind, flexible-dose, multicenter study. J Clin Psychiatry. 2008 Jan;69(1):106-13. doi: 10.4088/jcp.v69n0114. PMID 18312044
- [Derived] Keefe RS, Sweeney JA, Gu H, Hamer RM, Perkins DO, McEvoy JP, Lieberman JA. Effects of olanzapine, quetiapine, and risperidone on neurocognitive function in early psychosis: a randomized, double-blind 52-week comparison. Am J Psychiatry. 2007 Jul;164(7):1061-71. doi: 10.1176/ajp.2007.164.7.1061. PMID 17606658
- [Derived] McEvoy JP, Lieberman JA, Perkins DO, Hamer RM, Gu H, Lazarus A, Sweitzer D, Olexy C, Weiden P, Strakowski SD. Efficacy and tolerability of olanzapine, quetiapine, and risperidone in the treatment of early psychosis: a randomized, double-blind 52-week comparison. Am J Psychiatry. 2007 Jul;164(7):1050-60. doi: 10.1176/ajp.2007.164.7.1050. PMID 17606657